CLINICAL TRIAL: NCT04156997
Title: Extreme Lipids Repository
Status: Active, not recruiting | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Anand Rohatgi, Professor of Medicine, University of Texas Southwestern Medical Center
Other Study IDs: STU-2018-0429; 1K24HL146838-01 (NIH)
Record Dates: First submitted 2019-10-10; First posted 2019-11-08 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Lipoprotein Disorder
Keywords: Lipoproteins; Cholesterol; High Density Lipoproteins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Plasma, Serum, DNA, Cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with extreme lipid phenotypes: Adult patients (age 18 years or older) diagnosed with any lipid or metabolic disorder including hyperlipidemia, dyslipidemia, hyperlipoproteinemia, low HDL levels and deranged lipoprotein metabolism
  Interventions: Other: No intervention is involved in this study
- Healthy volunteers: Healthy adult volunteers with normal lipid metabolism will be recruited for the purpose of comparison
  Interventions: Other: No intervention is involved in this study

INTERVENTIONS:
Other: No intervention is involved in this study — No intervention is involved in this study

SUMMARY:
This is a prospective, observational study to establish a repository of samples from patients with extreme lipid phenotypes including but not limited to hyperlipidemia, dyslipidemia, hyperlipoproteinemia, extreme low/high HDL levels and deranged lipoprotein metabolism. The investigators plan to conduct sophisticated composition and functional analyses as well as genetic analysis to better understand the determinants of extreme lipid derangements.

DETAILED DESCRIPTION:
Participants will be recruited from clinical encounters within the University of Texas (UT) Southwestern Medical Center and Parkland Hospital by screening the Electronic Medical Record (EMR) for those with lipid labs and values that satisfy criteria for extreme values. Identified participants will be recruited to provide health information via survey, permission to extract clinical information from the EMR, and blood collection for future analyses. Measurements will span direct measurement of circulating species, genetic analyses, and analysis of circulating cells. The blood specimens will be stored for future studies and collaborations and thus, will constitute a blood-based repository. All study procedures are experimental but do not involve an actual intervention.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (age 18 years or older) diagnosed with any lipid or metabolic disorder including hyperlipidemia, dyslipidemia, hyperlipoproteinemia, low HDL levels and deranged lipoprotein metabolism

Exclusion Criteria:

* Anyone under 18 years of age will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with lipid and metabolism disorders and up to 50 healthy volunteers (age 18 years or older) with a normal lipid metabolism.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2019-05-10 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Biological sample collection for repository | Day 1
  Blood samples will be collected for preparation of plasma and serum, extraction of DNA and isolation of circulating cells. Future analysis include genomic, proteomic and metabolomic analysis
Data collection for repository | Day 1
  Demographic information, clinical history and lipid related bio-marker information will be collected from participants

CONTACTS AND LOCATIONS:
Overall Officials: Anand Rohatgi, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (2):
- United States (2):
  - Parkland Health Hospital System, Dallas, Texas
  - University of Texas Southwestern Medical Center - Ambulatory Clinic, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
Deidentified demographics, risk factors, clinical history, and research-based measures will be shared with other researchers with appropriate approval.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data will become available after completed enrollment of any participant. The data will be available for the duration of the registry.
Access Criteria: Researchers may request data from the PI, Dr. Anand Rohatgi. Once approval is given and appropriate regulatory approvals are in place, access may be granted and data shared.